CLINICAL TRIAL: NCT05451056
Title: An Open-label, Phase 2trial of Sotorasib in KRAS G12C-mutant Non-small-cell Lung Cancer(NSCLC) Patients and a Translational Study to Find Acquired Resistance Mechanism to Sotorasib
Acronym: breakthrough
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-1768
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sotorasib (Experimental): Sotorasib will be given 960mg daily PO until disease progression or unacceptable toxicity .
  Interventions: Drug: sotorasib

INTERVENTIONS:
Drug: sotorasib — Sotorasib will be given 960mg daily PO until disease progression or unacceptable toxicity.

SUMMARY:
Lung cancer is the most common type of cancer occurring in both males and females worldwide (WHO statistics, 2018), and the 5-year survival rate for advanced NSCLC is low (between 6% and 33%, depending on the stage. The rat sarcoma (RAS) proto-oncogene has been identified as an oncogenic driver of tumorigenesis in several cancers, including NSCLC. The RAS proteins can be mutationally activated at codons 12, 13, or 61, leading to human cancers. Different tumor types are associated with mutations in certain isoforms of RAS, with Kirsten rat sarcoma viral oncogene homolog (KRAS) being the most frequently mutated isoform in most cancers. While the role of KRAS mutations in human cancers has been known for decades, no anti-cancer therapies specifically targeting KRAS mutations have been successfully developed, largely because the protein has been intractable for inhibition by small molecules. AMG 510 is a small molecule that specifically and irreversibly inhibits the KRAS G12C mutated protein.

Nonclinical studies of AMG 510 have demonstrated inhibition of growth and regression of cells and tumors harboring KRAS p.G12C, and in clinical Study 20170543, AMG 510 demonstrated antitumor activity in KRAS p.G12C mutated NSCLC. These data suggest that inhibition of KRAS G12C may have therapeutic benefit for subjects with KRAS p.G12C driven cancers.

Recently development of liquid biopsy technology has enabled detection of KRAS-driven cancer with plasma ctDNA analysis. Therefore, in this study, we aim to conduct a phase 2 trial of sotorasib in KRAS G12C mutant-patients, and conduct pre-treatment and post-treatment biopsies using tissue and liquid to identify novel mechanisms of acquired resistance to sotorasib in these patients. Total sample size is 37 patients, Sotorasib will be given 960mg daily until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or subject's legally acceptable representative has provided informed consent prior to initiation of any study specific activities/procedures.
2. Age ≥19 years of age
3. Histologically or pathologically documented, locally-advanced and unresectable or metastatic NSCLC.
4. have documentation of KRAS p.G12C mutation confirmed by local testing through the current protocol or have documentation of KRAS p.G12C mutation prior to enrollment.
5. Subjects will have received and progressed or experienced disease recurrence on or after receiving at least 1 prior systemic therapy for locally advanced and unresectable or metastatic disease.
6. Adjuvant therapy will count as a line of therapy if the subject progressed on or within 6 months of adjuvant therapy administration.
7. In locally advanced and unresectable NSCLC, disease progression on or within 6 months of end of prior curatively intended multimodal therapy will count as a line of therapy. If chemoradiation is followed by planned systemic therapy without documented progression between chemoradiation and systemic therapy, the entire treatment course counts as one line of therapy.
8. Maintenance therapy following platinum doublet-based chemotherapy is not considered as a separate line of therapy.
9. Subjects must have archived tumor tissue samples (formalin fixed, paraffin embedded [FFPE] sample [FFPE of excisional, core needle, or fine needle aspirate] collected within 5 years) or be willing to undergo pre-treatment b iopsy (excisional, core needle, or fine needle aspirate) for tissue prior to enrollment.
10. Measurable disease per RECIST v1.1 criteria.
11. ECOG Performance Status of ≤ 1
12. Adequate hematologic laboratory assessments, defined as the following within 28 days prior to start of study therapy:

    1. Absolute neutrophil count (ANC) ≥ 1500 cells/μl (without granulocyte colony-stimulating factor support within 10 days of laboratory test used to determine eligibility)
    2. Hemoglobin ≥ 9.0 g/dL (without transfusion within 2 weeks of laboratory test used to determine eligibility)
    3. Platelet count ≥ 100,000/μl (without transfusion within 2 weeks of laboratory test used to determine eligibility)
13. Life expectancy of > 3 months, in the opinion of the investigator
14. Adequate liver function, defined as the following:

    1. Aspartate aminotransferase (AST) and, alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN), except if alkaline phosphatase > 2.5 times the ULN, then AST and/or ALT must be ≤ 1.5 times the ULN
    2. Serum bilirubin ≤ 1.0 x ULN
    3. International normalized ratio (INR) and activated partial thromboplastin time ≤ 1.5 x ULN
    4. Serum creatinine ≤1.5 x ULN OR creatinine clearance ≥ 60 mL/min. Cockcroft- Gault formula will be used for creatinine clearance calculation. Twenty-four hour urine collection is not required but is allowed.
15. QTc ≤ 470 msec in females and ≤ 450 msec in males (based on average of screening triplicates)

    -Subject should perform 12-lead ECG 3times within 15minutes at intervals of 2-5 minutes after resting in the sitting position for 5minutes.
16. Ability to take oral medications and willing to record daily adherence to investigational product

Exclusion Criteria:

1. Previously identified driver mutation (according to local standard of care or guidelines) other than KRAS p.G12C for which an approved therapy is available (including EGFR, ALK, ROS1, BRAF etc)
2. Active brain metastases. Subjects who have had brain metastases resected or have received whole brain radiation therapy ending at least 4 weeks (or stereotactic radiosurgery ending at least 2 weeks) prior to study day 1 are eligible if they meet all of the following criteria:

   1. residual neurological symptoms grade ≤ 2;
   2. on stable doses of dexamethasone or equivalent for at least 2 weeks, if applicable; and
   3. follow-up MRI performed within 30 days prior to enrollment shows no progression or new lesions appearing.
3. Leptomeningeal disease.
4. Exclusion of hepatitis infection based on the following results and/or criteria:

   1. Positive hepatitis B surface antigen (HepBsAg) (indicative of chronic Hepatitis B or recent acute hepatitis B)
   2. Subjects with a prior history of HBV proven to be positive for hepatitis B core antibody

      1. Surface antigen (HBsAg) is negative
      2. It is suitable if the HBV deoxyribonucleic acid (DNA; viral load) is less than the lower limit of quantitation according to the local test. Subjects positive for HBsAg due to recent vaccination are eligible if their HBV DNA (viral load) is below the lower limit of quantitation according to local testing.
5. Malignancy other than NSCLC within 2 years prior to first dose of drug, with the exception of those with a negligible risk of metastases or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal cell carcinoma, cutaneous squamous cell carcinoma, localized prostate cancer treated with curative intent, or ductal carcinoma in situ treated surgically with curative intent).
6. Significant gastrointestinal disorder that results in significant malabsorption, requirement for intravenous alimentation, or inability to take oral medication.
7. Significant cardiovascular disease, myocardial infarction within 6 months prior to study day 1, unstable arrhythmias or unstable angina.
8. Severe infections within 4 weeks prior to first dose of drug including, but not limited to hospitalization for complications of infection, bacteremia or severe pneumonia.
9. Subjects participating in other clinical trials are excluded.
10. Previous treatment with sotorasib or other KRAS G12C inhibitor
11. Female subjects of childbearing potential unwilling to use 1 highly effective method of contraception during treatment and for an additional 7 days after the last dose of sotorasib.
12. Female subjects of childbearing potential with a positive pregnancy test assessed at Screening or day 1 by a serum pregnancy test and/or urine pregnancy test.
13. Male subjects with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 7 days (sotorasib).
14. Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, Clinical Outcome Assessments) to the best of the subject and investigator's knowledge.
15. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of start of therapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  OS is measured from the date of start of study to the date of death from any cause.
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS is measured from the date of start of study to the date of disease progression or death from any cause.
Objective response rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  It is evaluated by taking CT of the chest and abdomen (including liver and adrenal glands) or MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Byoung Chul Cho, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No